

Kaushik Mukherjee MD MSCI FACS Associate Professor of Surgery Chief, Division of Acute Care Surgery Medical Director, Adult Level I Trauma Center 11175 Campus Street, CP 21111 Loma Linda, CA 92350

Phone: (909) 651-5948 Fax: (909) 558-0236 Email: kmukherjee@llu.edu

ClinicalTrials.Gov

July 17, 2025

Dear Sir or Madam,

This letter is intended to clarify the query as regards the study protocol date being 3/25/2021. The study protocol was not further amended during the course of the trial and this is the most recent version of the document.

Sincerely,

Kaushik Mukherjee MD MSCI FACS